CLINICAL TRIAL: NCT01518439
Title: Instrumental and Manual Increase of Couch in Neuromuscular Patients: Effects of Different Techniques on the Generated Flow
Brief Title: Instrumental and Manual Increase of Couch in Neuromuscular Patients
Acronym: OPTICOUGH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre d'Investigation Clinique et Technologique 805 (Other)
Collaborators: Adep Assistance (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011-A00879-32
Record Dates: First submitted 2012-01-11; First posted 2012-01-26 (Estimated); Last update posted 2013-07-19 (Estimated); Status verified 2013-07

CONDITIONS: Neuromuscular Disease; Chronic Respiratory Failure; Coughing
Keywords: neuromuscular; cough; restrictive
MeSH Terms: conditions — Neuromuscular Diseases; Cough | interventions — Physical Therapists

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- neuromuscular patients (Experimental): neuromuscular patients with cough inefficiency in a stable respiratory state upon inclusion
  Interventions: Device: Alpha 200®; Device: Alpha 200® + physiotherapist; Device: Cough Assist®; Device: Cough Assist® + physiotherapist; Other: physiotherapist

INTERVENTIONS:
Device: Alpha 200® — inspiratory capacity is increased with the use of constant pressure device: Alpha 200®
Device: Alpha 200® + physiotherapist — inspiratory capacity is increased with the use of constant pressure device (Alpha 200®) combined with the manual pressures techniques to increase cough by the physiotherapist
Device: Cough Assist® — increased inspiratory capacity and mechanical exsufflation with the use of insufflation-exsufflation device (Cough Assist®)
Device: Cough Assist® + physiotherapist — increased inspiratory capacity and mechanical exsufflation with the use of insufflation-exsufflation device (Cough Assist®) combined with the manual pressures techniques to increase cough by the physiotherapist
Other: physiotherapist — manual pressures techniques to increase cough applied by the physiotherapist

SUMMARY:
Inefficient cough is responsible of respiratory complications in neuromuscular patients which can lead to hospitalisation and can be life threatening. Techniques enhancing cough efficiency are successful in improving the clearance of bronchial secretions and help non invasive ventilation efficiency especially in case of acute respiratory failure. Combining mechanical exsufflation to the manual techniques of physiotherapy might enhance efficiency. Therefore the investigators want to compare cough efficiency under different techniques of instrumental and manual of cough assistance in order to determine the best combination to optimize cough flow.

DETAILED DESCRIPTION:
Hypothesis: Cough inefficiency in neuromuscular patients increases morbidity and mortality in case of airway infections and may lead to invasive ventilation. The use of techniques enhancing cough have been successful in improving the success of non invasive ventilation. We want to determine whether adding manual physiotherapist techniques to mechanical exsufflation improve cough efficiency and its ability to clear bronchial secretions.

Objectives: To compare cough flows obtained with different combination of the use of increased inspiratory capacity technique, mechanical insufflation-exsufflation technique and manually applied pressures techniques.

Method:open monocentric cross-over study (the patients are their own controls). Five combinations of cough increase techniques are compared Inclusion criteria: adult neuromuscular patients with a cough inefficiency at a stable state upon inclusion.

As this is a pilot study, 20 patients from the home ventilation unit of the intensive care of the Raymond Poincare teaching hospital (Garches, France) will be included during the usual follow-up of chronic respiratory failure.

ELIGIBILITY:
Inclusion Criteria:

* adult patients
* neuromuscular disorders with a respiratory restrictive syndrome (VC < 40% and/or cough flow < 180 L/min and/or Pe max < 40 cmH2O)
* non invasive ventilation
* stable respiratory state > 1 month before inclusion
* signed informed consent form

Exclusion Criteria:

* unstable respiratory state with increased bronchial secretions
* unstable hemodynamics
* pneumothorax and or emphysema
* tracheostomy
* major bulbar involvement with swallowing dysfunction with the liquids
* Persons under Guardianship or Trusteeship
* Pregnant women
* not covered by the social security system
* refusal of study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-01; Primary Completion 2012-01 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
cough flow obtained from the combination of mechanical and manual cough assistance techniques | 2 Hours

SECONDARY OUTCOMES:
duration of efficient cough flow (above 180 l/min)under each cough assistance technique | 2 Hours
respiratory comfort | 2 Hours
  evaluation with a visual analogical scale
subjective evaluation of cough efficiency | 2 Hours
  evaluation with a visual analogical scale
Respiratory comfort | 2 Hours
  evaluation with the Borg dyspnea scale

CONTACTS AND LOCATIONS:
Overall Officials: Frederic Lofaso, Md-PhD, Study Director — University of Versailles; Helene Prigent, MD-PhD, Principal Investigator — University of Versailles
Locations (1):
- RAYMOND POINCARE Hospital, Garches, Garches, France

REFERENCES:
- [Derived] Morrow B, Argent A, Zampoli M, Human A, Corten L, Toussaint M. Cough augmentation techniques for people with chronic neuromuscular disorders. Cochrane Database Syst Rev. 2021 Apr 22;4(4):CD013170. doi: 10.1002/14651858.CD013170.pub2. PMID 33887060